CLINICAL TRIAL: NCT03977142
Title: Accuracy of the Noninvasive Radical-7 Pulse Co-oximeter at Detecting Hemoglobin Changes in Pediatric Cardiac Intensive Care
Brief Title: Validity of Radical 7 Masimo Monitor at Measuring Hemoglobin in Pediatric Cardiac Intensive Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Genevieve Du Pont-Thibodeau, Pediatric Intensivist, St. Justine's Hospital
Other Study IDs: HgPCICU
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Evaluate the Accuracy of the Masimo Radical 7 Hemoglobin Noninvasive Monitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Radical 7 Masimo Hemoglobin pulse co-oximeter non invasive monitor — Measure hemoglobin levels non invasively by pulse co-oximeter

SUMMARY:
Fifty percent of children that survive a critical illness are anemic at discharge from the pediatric intensive care unit (PICU)(1). Given that there are approximately 9000 PICU admissions/year in Canada, this represents almost 4500 children per year. Anemia is associated with abnormal neurocognitive development in infants and young children. A contributor to PICU anemia is the excessive amount of blood testing and iatrogenic blood losses(2). Non-invasive continuous hemoglobin monitoring (Sp-Hb) have been developed in the medical setting in an attempt to minimize invasive blood testing and reduce blood losses. The Radical 7 Masimo device (Masimo corporation, Irvine, CA) is one of the popular devices used for non-invasive hemoglobin monitoring. Its accuracy has been previously investigated in various populations(3-6). The objective of this study is to investigate the validity of the Radical 7 Masimo device at measuring hemoglobin trends non-invasively in critically ill children.

DETAILED DESCRIPTION:
This will be a prospective observational study. We will include 1) all patients that are admitted to the PICU of the CHUSJ after a cardiac surgery, 2) that are aged less than 6 months on the day of admission and that 3) have an arterial line inserted.

All children studied will have an arterial line inserted at the time of surgery that will allow for arterial-Hb measurements. As this study is strictly observational, all arterial-Hb measurements will be requested by the medical treating team as clinically indicated. We will install, on admission, the spectrophotometric adhesive sensor required for Sp-Hb measurements on each patient (Masimo Rainbow R1 20 for children over 30 kg and R1 20L for those under 30 kg). The sensor will be applied on the hand or foot that does not have an arterial cannula. The sensor will be covered with an impermeable black shield to prevent optical interference.

We will collect all the arterial-Hb measurements performed in the 48 hours after PICU admission as well as all the Sp-Hb readings performed at the time of the arterial samples. The blood samples drawn from the arterial catheter will be analyzed using a laboratory CO-oximeter (model ABL820; Radiometer, Copenhagen, Denmark). Simultaneous recording of Sp-Hb will performed within 10 seconds after the arterial blood sample is drawn. We will also collect demographic data and clinical data on each patient; age, weight, sex, ethnicity, type of cardiac surgery, blood transfusions. At the CHUSJ PICU, all clinical and demographic data is systematically recorded in our electronic database (Intellispace Critical Care and Anesthesia, Philips Medical Systems). Data on red cell transfusions are recorded through the TracelineTM database that is made available to our research group through Héma-Québec. Data will be extracted from our database by our research assistant.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients that are admitted to the PICU of the CHUSJ after a cardiac surgery, 2) that are aged less than 6 months on the day of admission and that 3) have an arterial line inserted.

Max Age: 6 Months | Sex: All
Age Groups: Child
Study Population: Children admitted to the PICU after a cardiac surgery
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
To determine the precision of the Radical-7 pulse co-oximeter at detecting changes in Hb levels when comparted to arterial-Hb levels changes in children admitted to the PICU after a cardiac surgery. | 3 months
To determine the precision of the Radical-7 pulse co-oximeter at measuring Hb values when compared to arterial-Hb in children admitted to the PICU after a cardiac surgery. | 3 months

IPD SHARING:
Plan to Share IPD: No